CLINICAL TRIAL: NCT05500404
Title: Diagnostic Accuracy of Placental Thickness in Lower Uterine Segment Measured By Ultrasound in Prediction of Placenta Accreta Spectrum in Patients With Placenta Previa. A Diagnostic Test Accuracy Study
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer, Ain Shams Maternity Hospital
Other Study IDs: 5
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cases with morbidly adherent placenta who will undergo cesarean hysterectomy will have thier uteri sent for histopathologic examination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound measurment of placental thickness — The maximum placental thickness in the lower uterine segment will obtained using trans-abdominal ultrasound scan. For the image to be deemed suitable, a midline sagittal section of the lower uterine segment (with the implanted placenta) and the cervical canal, with the intervening urinary bladder will be required (Bhide et al., 2019). The measurement will be performed by a researcher who will be blinded to the final diagnosis.

SUMMARY:
Current prenatal diagnosis of placenta accrete spectrum disorders relies on subjective individual interpretations of visual sonographic findings on grayscale and color Doppler imaging. When blinded to clinical data, there is significant interobserver variability in the diagnosis of invasive placentation.

This study will evaluate placental thickness among pregnant women with placenta previa and determine if increased placenta thickness correlates with the risk for placenta accreta spectrum (PAS) disorders.

DETAILED DESCRIPTION:
Placenta accreta spectrum is one of the most dangerous conditions associated with pregnancy, because hemorrhage may result in multisystem organ failure, disseminated intravascular coagulation, need for admission to an intensive care unit, hysterectomy, and even death. The reported incidence of placenta accrete spectrum disorder has increased over time and is currently between 1 in 533 to 1 in 300 pregnancies. Prior cesarean delivery and especially multiple cesarean deliveries are major risk factors. The spectrum includes placenta accreta (attachment of the placenta to myometrium without intervening decidua), placenta increta (invasion of the trophoblast into the myometrium), and placenta percreta (invasion through the myometrium, serosa, and into surrounding structures). PAS is linked to placenta previa, and there is a lot of overlap in imaging findings between the two processes. PAS problems affect approximately 11% of people with placenta previa. Differentiating between placenta previa with and without PAS problems is crucial in clinical practice. A finding of placenta previa together with a history of cesarean delivery has long been an indication for counseling patients on their risk of PAS in a current pregnancy, as the risk for placenta accreta in the presence of placenta previa increases with each subsequent cesarean delivery. Aside from cesarean deliveries and placenta previa, other risk factors have been identified for PAS, including past uterine surgeries, in vitro fertilization (IVF), multiparity, maternal age, and even female sex of the infant. Prenatal diagnosis of AIP has been shown to reduce maternal morbidity associated with this condition, most likely due to the opportunity to plan management in advance. Ultrasound is the primary investigation for prenatal diagnosis of morbidly adherent placenta, and the diagnostic accuracy is good both in retrospective, as well as prospective case series. Placental localization with transabdominal sonography (TAS) has been a standard practice for a long time. Despite its availability and noninvasive nature, accuracy of TAS may be limited by many factors, such as the posterior implantation of placenta, being obscured by the fetal head, an under-filled or over-distended bladder, and presence of blood clots, fibroids, uterine contractions, and obesity. These limitations are overcome by transvaginal sonography (TVS), which provides a better resolution by using a higher frequency transducer, shorter distance from the transducer to the internal os, and is not affected by the over- or under-filling of the bladder. Although ultrasonography's sensitivity and specificity for detecting accreta have been reported to be excellent, ranging from 80 to 90%, there was considerable difference among "experts" in predicting whether PAS was present. With placental implantation into the cesarean section scar, the center of the placental disc would be in the vicinity of the lower uterine scar. If placental implantation was near the scar but not in it, only the thinner placental margin might encroach into the lower uterine segment. The investigators therefore hypothesized that the placenta is thicker with AIP in women with a low-lying placenta or placenta previa. So, the investigators hypothesize that placental thickness will be directly related to placental invasion in cases of placenta accrete spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with ultrasound diagnosis of placenta previa or low lying placenta
* Gestational age above 26 weeks
* singleton pregnancy
* fetal life positive
* Past history of cesarean section regardless of the number

Exclusion Criteria:

* Hemodynamically unstable women.
* Patients with pregestational or gestational DM.
* Multiple gestation.
* Medical disorders which can lead to uteroplacental insufficiency (preeclampsia - SLE - antiphospholipid antibody syndrome).
* Any condition which can lead to enlarged placenta such as fetal hydrops

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with placenta Previa attending outpatient obstetric clinic at Ain Shams University Maternity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Placental thickness threshold | after 26 weeks of pregnancy
  Threshold of placental thickness which can be used as cutoff level with appropriate sensitivity and specificity so it can be used as a screening test for such morbid condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mamdouh, MD, Study Director — Ainshams university maternity hospital
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silver RM, Branch DW. Placenta Accreta Spectrum. N Engl J Med. 2018 Apr 19;378(16):1529-1536. doi: 10.1056/NEJMcp1709324. No abstract available. PMID 29669225
- [Background] Li Y, Choi HH, Goldstein R, Poder L, Jha P. Placental thickness correlates with placenta accreta spectrum (PAS) disorder in women with placenta previa. Abdom Radiol (NY). 2021 Jun;46(6):2722-2728. doi: 10.1007/s00261-020-02894-9. Epub 2021 Jan 2. PMID 33388802
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Morgan EA, Sidebottom A, Vacquier M, Wunderlich W, Loichinger M. The effect of placental location in cases of placenta accreta spectrum. Am J Obstet Gynecol. 2019 Oct;221(4):357.e1-357.e5. doi: 10.1016/j.ajog.2019.07.028. Epub 2019 Jul 22. PMID 31344349
- [Background] Bhide A, Laoreti A, Kaelin Agten A, Papageorghiou A, Khalil A, Uprichard J, Thilaganathan B, Chandraharan E. Lower uterine segment placental thickness in women with abnormally invasive placenta. Acta Obstet Gynecol Scand. 2019 Jan;98(1):95-100. doi: 10.1111/aogs.13422. Epub 2018 Aug 2. PMID 29978457
- [Background] Petpichetchian C, Pranpanus S, Suntharasaj T, Kor-Anantakul O, Hanprasertpong T. Comparison of transabdominal and transvaginal sonography in the diagnosis of placenta previa. J Clin Ultrasound. 2018 Jul;46(6):386-390. doi: 10.1002/jcu.22600. Epub 2018 Apr 25. PMID 29693718
- [Derived] Elmaraghy AM, Taha Fayed S, Abd ElHamid Ali M, Ali Hassanien M, Mohamed Mamdouh A. Diagnostic Accuracy of Placental Thickness in Lower Uterine Segment Measured by Ultrasound in Prediction of Placenta Accreta Spectrum in Patients with Placenta Previa. A Diagnostic Test Accuracy Study. Int J Womens Health. 2023 Feb 16;15:311-320. doi: 10.2147/IJWH.S399520. eCollection 2023. PMID 36814526